CLINICAL TRIAL: NCT01833897
Title: NMDA Antagonists in Bipolar Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6535
Record Dates: First submitted 2013-04-12; First posted 2013-04-17 (Estimated); Results first posted 2016-06-01 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-03

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Standard of Care; Quetiapine Fumarate; Olanzapine; Fluoxetine; Ketamine; Cycloserine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ketamine and DCS treatment (Experimental): Standard of Care: Subjects will receive treatment with either quetiapine, olanzapine-fluoxetine, or lurasidone. If after about 2 week, subjects are symptomatic, subjects will receive infusion of ketamine hydrochloride (0.5 mg/kg). After the ketamine phase, subject who show improvement will begin an 8-week treatment of oral D-cycloserine.
  Interventions: Drug: Standard of Care; Drug: Ketamine; Drug: D-cycloserine

INTERVENTIONS:
Drug: Standard of Care — Quetiapine, olanzapine-fluoxetine, and lurasidone are approved treatments for bipolar depression. Quetiapine dosing will follow the product label(Anon), and will be titrated over the first 4 days to the target dose of 300 mg. Olanzapine-fluoxetine dosing will also follow standard guidelines. Lurasidone will be started at 20 mg, and titrated up to 60 mg daily as clinically indicated. Study physicians will use clinical judgment to choose between standard-of care treatments, and have the option to titrate standard-of-care within approved ranges, and to prescribe adjunctive benztropine and benzodiazepines if clinically indicated.
  Other Names: Quetiapine; Olanzapine; fluoxetine
Drug: Ketamine — Ketamine administration will be carried out according to the methods as described by previous studies. Subjects will receive ketamine hydrochloride (0.5 mg/kg) intravenously during 40 minutes. This dosage was selected based on previous trials of ketamine for the treatment of refractory depression and bipolar depression. Vital signs (blood pressure, heart rate) will be closely monitored throughout the time of infusion. Subjects will be evaluated for 2 consecutive days during this phase; i.e. treatment days (day 1) and rating days (day 2). Non-responders to ketamine will not proceed into the DCS phase. Response will be a 25% improvement on the Hamilton Depression Rating Scale (HDRS).
  Other Names: Ketamine Hydrochloride
Drug: D-cycloserine — Immediately after the ketamine infusion, subjects will begin an eight-week treatment of DCS adjunctive to standard of care. DCS dosing will begin at 250 mg for three days→500mg (2 capsules)/day for 1 week → 750 mg (3 capsules)/day for 1 week → and 1000 mg (4 capsules)/day for the remainder of the study.
  Other Names: DCS

SUMMARY:
The purpose of this study is to test whether ketamine and D-cycloserine can be safely and effectively used for the treatment of depression. The investigators hypothesize that ketamine will serve as a rapid acting and safe antidepressant in patients with bipolar depression, and furthermore, that D-cycloserine will serve as an effective therapy following ketamine treatment.

DETAILED DESCRIPTION:
Bipolar disorder affects 2% of the population in the United States and the depressive phase contributes disproportionally to morbidity and mortality. At present, few approved treatments for bipolar depression are available, and have primarily depended on manipulations of brain monoaminergic systems. In contrast, recent studies suggest that the N-methyl-D-aspartate glutamate-receptor (NMDAR) antagonist, ketamine, may provide near-immediate relief for treatment resistant depression. Its utility during long-term treatment, however, is limited by its psychotomimetic potency and the need for repeated IV infusions. D-cycloserine (DCS) is an approved oral antibiotic for tuberculosis drug and a well-studied mixed agonist/antagonist at the NMDAR/glycine binding site. DCS showed preliminary evidence of efficacy in a pilot study. DCS would thus be practical from both a safety and route of administration perspective. The present study will explore the feasibility and safety of DCS for maintenance treatments, as measured by magnetic resonance spectroscopy (MRS).

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with Diagnostic and Statistical Manual, Version 4 (DSM-IV) diagnosis of bipolar disorder I or II, current major depressive episode without psychotic features, 18-60
* Insufficient therapeutic response during the current episode
* Medically stable for study participation
* Judged clinically not to be at significant suicide or violence risk
* Subject is off all psychotropic and other types of drugs likely to interact with glutamate for at least 14 days before starting the study. One exception is chloral hydrate or short acting benzodiazepines for distressing anxiety or insomnia (up to 72 hours prior to each MRI scan). In addition, subjects will be off antipsychotics for 1 month and off fluoxetine for 6 weeks prior to the study.
* Subject is likely to be able to tolerate a medication washout. Only subjects who have failed their current medication regiment will be washed off medications.

Exclusion Criteria:

* History of chronic psychosis or drug induced psychosis of any kind
* Current DSM-IV diagnosis of drug abuse/dependence in the last six months. Subjects must have a negative drug screen at baseline.
* Women will be excluded if they are pregnant lactating, or not either surgically-sterile or using appropriate methods of birth control. Women must agree to continue using applicable birth control throughout the trial. All women of child-bearing potential must have a negative urine pregnancy test
* Taking any medication contraindicated with ketamine or DCS (ethionamide, isoniazid)
* History of seizures, renal insufficiency or congestive heart failure
* History of clinically significant violence
* History of ketamine abuse/dependence or prior clinically significant adverse reaction to ketamine
* Current alcohol abuse or dependence
* Untreated hypertension
* Clinically abnormal liver function tests (LFTs), thyroid, renal function or anemia
* Metal implants, pacemaker, other metal (e.g. shrapnel or surgical prostheses) or paramagnetic objects contained within the body which may present a risk to the subject or interfere with the MR scan.
* Medicinal patch, unless removed prior to the MR scan

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2013-03; Primary Completion 2014-07 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua T Kantrowitz, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ketamine and DCS Treatment
Started | 8
Completed | 7
Not Completed | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ketamine and DCS Treatment
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 3
Montgomery Asberg Depression Rating scale [Mean (Standard Deviation); unit: units on a scale] — Measure of depression: Higher MADRS score indicates more severe depression, and each item yields a score of 0 to 6. The overall score ranges from 0 to 60
  units on a scale | 29 (6)
Hamilton Depression Rating Scale (HAM-D) [Mean (Standard Deviation); unit: units on a scale] — Depression rating scale: Range 0-53, higher scores indicate worse depression.
  0-7 = Normal 8-13 = Mild Depression 14-18 = Moderate Depression 19-22 = Severe Depression
  ≥ 23 = Very Severe Depression
  units on a scale | 18.8 (6.7)
Hamilton Depression Rating Scale (HAM-D) suicide item [Mean (Standard Deviation); unit: units on a scale] — Item 3 of scale (range 0-4) with higher scores indicating higher symptoms
  units on a scale | 1.25 (0.9)
Loss of Motivated Behavior HAM-D Factor [Mean (Standard Deviation); unit: units on a scale] — Includes the total of four HAM-D items: (Item 7: Work and activities, Item 12. Somatic symptoms (appetite), Item 14. Genital symptoms (libido), and Item 16. Weight loss). Range 0-11, higher scores indicate worse symptoms.
  units on a scale | 5 (1.6)
Hamilton Anxiety Rating Scale (HAM-A) [Mean (Standard Deviation); unit: units on a scale] — Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indi- cates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
  units on a scale | 12.6 (4.2)
Beck's depression inventory [Mean (Standard Deviation); unit: units on a scale] — Ranges from 0-63, with Higher total scores indicate more severe depressive symptoms.
  The standardized cutoffs used:
  0-13: minimal depression 14-19: mild depression 20-28: moderate depression 29-63: severe depression.
  units on a scale | 31.4 (10.4)
Time of treatment resistance [Mean (Standard Deviation); unit: Months] | 3.3 (4)

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Depression Rating Scale (HAM-D)
Description: Depression rating scale: Range 0-53, higher scores indicate worse depression. 0-7 = Normal 8-13 = Mild Depression 14-18 = Moderate Depression 19-22 = Severe Depression
  ≥ 23 = Very Severe Depression
Time Frame: 8 weeks
Population: bipolar depression
Measure: Mean (Standard Deviation); unit: units on a scale (final score)
Arm/Group | Ketamine and DCS Treatment
Number analyzed (Participants) | 8
units on a scale (final score) | 9.5 (7)
Statistical Analysis 1: Comparison: Ketamine and DCS Treatment; Test type: Superiority or Other; p < 0.001, linear mixed model — F1,6.4=161.8,

2. Secondary Outcome: Loss of Motivated Behavior HAM-D Factor
Description: includes the total of four HAM-D items: (Item 7: Work and activities, Item 12. Somatic symptoms (appetite), Item 14. Genital symptoms (libido), and Item 16. Weight loss). Range 0-11, higher scores indicate worse symptoms
Time Frame: 8 weeks
Population: bipolar depression
Measure: Mean (Standard Deviation); unit: units on a scale (final score)
Arm/Group | Ketamine and DCS Treatment
Number analyzed (Participants) | 8
units on a scale (final score) | 1.6 (1.9)
Statistical Analysis 1: Comparison: Ketamine and DCS Treatment; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis

3. Secondary Outcome: HAM-D Suicide Item
Description: Ham-D suicide item: range 0-4, higher scores indicate worse symptoms
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale (final)
Arm/Group | Ketamine and DCS Treatment
Number analyzed (Participants) | 8
units on a scale (final) | 0.3 (0.5)
Statistical Analysis 1: Comparison: Ketamine and DCS Treatment; Test type: Superiority or Other; p = 0.026, ANOVA

4. Secondary Outcome: Hamilton Anxiety Scale
Description: Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indi- cates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale (final score)
Arm/Group | Ketamine and DCS Treatment
Number analyzed (Participants) | 8
units on a scale (final score) | 6.4 (5)
Statistical Analysis 1: Comparison: Ketamine and DCS Treatment; Test type: Superiority or Other; p = 0.011, ANOVA

5. Secondary Outcome: Beck's Depression Inventory
Description: Range 0-63, with higher scores worse. Total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale (final score)
Arm/Group | Ketamine and DCS Treatment
Number analyzed (Participants) | 8
units on a scale (final score) | 10.8 (9.2)
Statistical Analysis 1: Comparison: Ketamine and DCS Treatment; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis

ADVERSE EVENTS:
Arm/Group | Ketamine and DCS Treatment
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 4/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine and DCS Treatment (N=8)
headache (Nervous system disorders) | 2 (2) — mild
sedation (Nervous system disorders) | 3 (3) — mild
phosphenes (Eye disorders) | 1 (1)
hypomania (Psychiatric disorders) | 1 (1) — after stopping clinical medications

LIMITATIONS AND CAVEATS:
Limitations include the small-sample and a non-placebo controlled, open-label design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No